CLINICAL TRIAL: NCT01466192
Title: A Phase 3 Study of MP-424 in Combination With Peginterferon Alfa-2b and Ribavirin in Subjects With Genotype 2 Hepatitis C, Who Relapsed After Previous Treatment
Brief Title: Efficacy and Safety of MP-424, Peginterferon Alfa-2b and Ribavirin in Relapser Genotype 2 Hepatitis C Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060-A10
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis C
Keywords: Genotype 2
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP-424 (Experimental)
  Interventions: Drug: MP-424 (generic name:Telaprevir); Drug: Ribavirin; Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: MP-424 (generic name:Telaprevir) — 750mg q8h for 12 weeks
Drug: Ribavirin — 400 - 1000 mg/day based on body weight for 24 weeks
Drug: Peginterferon alfa-2b — 1.5mcg/kg/week for 24 weeks

SUMMARY:
This study will evaluate the efficacy and safety of MP-424 with Peginterferon Alfa-2b and Ribavirin (RBV) in patients with genotype 2 hepatitis C, who relapsed after previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 2, chronic hepatitis C
* Relapsers (patient who relapsed after previous treatment)
* Able and willing to follow contraception requirements

Exclusion Criteria:

* Cirrhosis of the liver or hepatic failure
* Hepatitis B surface antigen-positive or HIV antibodies-positive
* History of, or concurrent hepatocellular carcinoma
* History of, or concurrent depression, schizophrenia,; or suicide attempt in the past
* Pregnant, lactating, or suspected pregnant patients, or male patients whose female partner is pregnant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Toranomon Hospital, Minato-ku, Tokyo, Japan

REFERENCES:
- [Result] Kumada H, Sato K, Takehara T, Nakamuta M, Ishigami M, Chayama K, Toyota J, Suzuki F, Nakayasu Y, Ochi M, Yamada I, Okanoue T. Efficacy of telaprevir-based therapy for difficult-to-treat patients with genotype 2 chronic hepatitis C in Japan. Hepatol Res. 2015 Jul;45(7):745-54. doi: 10.1111/hepr.12416. Epub 2014 Nov 18. PMID 25196718

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP-424
Started | 108
Completed | 104
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | MP-424
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 53

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV RNA at 24 Weeks After Completion of Drug Administration (SVR, Sustained Viral Response)
Time Frame: After 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR
Arm/Group | MP-424
Number analyzed (Participants) | 108
percentage of subjects achieving SVR | 88.0 [80.3 to 93.4]

ADVERSE EVENTS:
Arm/Group | MP-424
Serious Adverse Events (participants affected / at risk) | 12/108
Other Adverse Events (participants affected / at risk) | 108/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=108)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Malaise (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=108)
Nasopharyngitis (Infections and infestations) | 42
Anaemia (Blood and lymphatic system disorders) | 86
Decreased appetite (Metabolism and nutrition disorders) | 54
Hyperuricaemia (Metabolism and nutrition disorders) | 28
Hypokalaemia (Metabolism and nutrition disorders) | 6
Insomnia (Psychiatric disorders) | 25
Headache (Nervous system disorders) | 48
Dysgeusia (Nervous system disorders) | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Nausea (Gastrointestinal disorders) | 43
Abdominal discomfort (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 28
Diarrhoea (Gastrointestinal disorders) | 21
Stomatitis (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 15
Cheilitis (Gastrointestinal disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 42
Alopecia (Skin and subcutaneous tissue disorders) | 33
Drug eruption (Skin and subcutaneous tissue disorders) | 25
Pruritus (Skin and subcutaneous tissue disorders) | 16
Eczema (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 26
Back pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pyrexia (General disorders) | 86
Malaise (General disorders) | 71
Injection site erythema (General disorders) | 30
Injection site reaction (General disorders) | 24
Influenza like illness (General disorders) | 7
Thirst (General disorders) | 6
White blood cell count decreased (Investigations) | 68
Platelet count decreased (Investigations) | 61
Blood creatinine increased (Investigations) | 40
Blood uric acid increased (Investigations) | 39
Hyaluronic acid increased (Investigations) | 23
Blood triglycerides increased (Investigations) | 18
Blood bilirubin increased (Investigations) | 17
Blood potassium decreased (Investigations) | 9
Blood phosphorus decreased (Investigations) | 9
Haemoglobin decreased (Investigations) | 8
Alanine aminotransferase increased (Investigations) | 6
Gamma-glutamyltransferase increased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other